CLINICAL TRIAL: NCT07038421
Title: The Investigation of Lower Extremity Problems, Gait and Falling Risk in Patient With Stroke
Brief Title: Gait and Falling Risk in Patient With Stroke
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-01/1115
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Gait; Proprioception

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stroke group: Individuals diagnosed with stroke at least 3 months ago by a neurologist
  Interventions: Other: Cognitive level; Other: Gait; Other: Spasticity; Other: Position sense; Other: Plantar sense

INTERVENTIONS:
Other: Cognitive level — The cognitive function was assessed with the Montreal Cognitive Assessment (MOCA). The total score ranges from 0 to 30, and scores of 21 and above indicate normal cognitive status
Other: Gait — The Dynamic Gait Index (DGI) was assessed for gait. The maximum total score is 24, with a lower DGI score indicating greater impairment in functional mobility and gait
Other: Spasticity — Spasticity was assessed using the Modified Ashworth Scale (MAS). In the MAS, muscles were recorded as 0, 1, 1, 1+, 2, 3, and 4 according to the resistance they gave to passive movement.
Other: Position sense — The position sense was measured using a dual digital inclinometer. The mean absolute error from three trials was recorded. As the mean absolute error increased, position sense deteriorated.
Other: Plantar sense — Plantar sensation was evaluated with the Semmes-Weinstein monofilament test (SWMT). The smallest monofilament value felt and correctly identified was recorded as the patient's threshold for light touch and pressure sensation. As the value increases, the underfloor sensation worsens.

SUMMARY:
This study focuses on the impact of lower extremity dysfunctions following stroke-such as muscle weakness, spasticity, and sensory impairments-on gait and fall risk. Post-stroke gait is typically slow, asymmetric, and functionally limited due to motor and sensory deficits. Spasticity, particularly in the lower limb muscles like the gastrocnemius, further complicates walking. Sensory issues, including reduced plantar sensation and joint position sense, also contribute to impaired mobility and balance. The study aims to examine the relationship between gait, plantar sensation, knee position sense, and spasticity, and how these factors influence fall risk in stroke patients.

The aim of the study is to investigate the relationship between gait and plantar sensation, knee position sensation, and spasticity based on these results. Another aim is to determine the effects of plantar sensation, knee position sensation, and spasticity on fall risk. We previously hypothesized that there is a relationship between gait and spasticity, position sense, plantar sensation. This study further hypothesizes hypothesises that parameters associated with gait will influence the risk of falls in patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with stroke by a specialist neurologist at least 3 months prior to the study
* Aged 18 years or older
* Having a cognitive level of above 21 points on the Montreal Cognitive Assessment (MoCA)
* Able to walk independently, with or without an assistive device
* Volunteering

Exclusion Criteria:

* Had any additional neurological disorder other than stroke
* Had a history of surgical intervention involving the lower extremities
* Had an orthopedic or rheumatologic condition affecting the lower extremities.

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Stroke patients
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Gait ability | one hour
  The Dynamic Gait Index (DGI) was developed to assess functional stability during gait. The lower score indicating greater impairment in gait. According to the DGI score, the cutoff value for fall risk was 16.5.

SECONDARY OUTCOMES:
Spasticity | One hour
  Spasticity was assessed using the MAS. As the MAS score increases, the severity of spasticity increases.
Position sense | one hour
  The knee position sense (60 degree) was measured using a dual digital inclinometer. An increase in the mean absolute error indicates that position sense is impaired.
Plantar sense | one hour
  Plantar sensation was evaluated with the monofilament test. As the monofilament value increases, sensation deteriorates.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Eyalet/Yerleşke, Turkey (Türkiye)